CLINICAL TRIAL: NCT03390920
Title: Evaluation of Regenerative Medicine Outcomes With Umbilical Allograft for Musculoskeletal Conditions
Brief Title: Evaluation of Outcomes With Umbilical Cord Allograft for Musculoskeletal Conditions Musculoskeletal Conditions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: R3 Stem Cell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2017/05/6
Record Dates: First submitted 2017-12-19; First posted 2018-01-04 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis; Tendinitis; Sports Injury; Degenerative Disc Disease; Degenerative Arthritis; Ligament Injury; Neuropathy; Pelvic Pain
Keywords: regenerative medicine; arthritis; amniotic; stem cell; growth factor; cartilage
MeSH Terms: conditions — Osteoarthritis; Tendinopathy; Athletic Injuries; Intervertebral Disc Degeneration; Pelvic Pain; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Umbilical Allograft (Experimental): The study is nonrandomized with one arm. Depending on the body area being treated, the amount of the product utilized will be either 1.0cc's or 2cc's.
  Interventions: Other: Umbilical Allograft

INTERVENTIONS:
Other: Umbilical Allograft — The umbilical allograft is regulated by the FDA and comes from a lab that is FDA registered.

SUMMARY:
The aim of the study is to determine the efficacy of an Amniotic Fluid Tissue Product for pain relief and functional improvements for all types of musculoskeletal conditions. The study is prospective, with outcome measures being obtained at numerous time points after the regenerative procedure.

DETAILED DESCRIPTION:
Medical providers are often faced with patients whose source of pain may be the result of an inflammatory response caused by trauma or disease. By managing the patient's inflammation, the clinician may see improved response to traditional pain management therapy and existing protocols.

Also, degenerative arthritis of spinal and extremity joints may lead to significant low back, knee, hip, shoulder pain etc, as the ratio of cartilage degradation to cartilage formation increases with age. An amniotic tissue derived product may prove to be an ideal non-steroidal and potentially regenerative therapy for use by the medical provider due to its unique characteristics.

The orthopedic application of amniotic fluid dates back to at least the 1930's. The placental membranes produce an array of immunosuppressive and anti-inflammatory molecules, which make these tissues suitable for use as a wound covering [or as an anti-inflammatory] in a clinical setting. In addition to structural properties, placental membrane and amniotic fluid (AF) is a rich source of growth factors, including organic compounds and nutrients, hyaluronic acids, amino acids, antioxidants and stem cells.

AF's anti-inflammatory actions may be mediated in part by its secretion of anti-inflammatory cytokines including interleukin-10, inhibin, activin, and interleukin-1 receptor antagonist as well as anti-inflammatory protease inhibitors such as ∞-1 anti-trypsin inhibitor and inter-a-trypsin inhibitor. AF may modulate acquired immunity by suppressing alloreactive responses and down regulating production of Th1 and Th2 cytokines.

In addition to having known anti-inflammatory qualities, placental membrane cells, derived from the layer of trophoblast cells covering the developing embryo, do not express MHC Class II antigens, which are responsible for the rapid rejection of allografts in humans. Because AF is immune privileged, it is an ideal allograft with no known graft-versus-host disease (GVHD).

The amniotic fluid product may provide not only an anti-inflammatory response, but also potentially yield regenerative effect or reduce further cartilage degeneration.

The objective of this study is to evaluate an amniotic fluid tissue product in the treatment of pain due to all types of musculoskeletal conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over.
2. Ability to attend follow up visits or at least converse on phone or complete email follow up forms.

4) Competent to understand the study protocol and provide voluntary informed consent.

Exclusion Criteria:

1. Active Infection
2. Pregnancy, Lactating
3. Clotting disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Short Musculoskeletal Function Assessment Questionnaire (SMFA) | Baseline and then Assess Changes Post Intervention at 4 weeks, 3 mths, 6 mths, 9 mths and one year
  The Short Musculoskeletal Function Assessment Questionnaire (SMFA) is designed to measure the functional status of patients with a broad range of musculoskeletal injuries and disorders.

SECONDARY OUTCOMES:
Work Status | Baseline and then Assess Changes Post Intervention at 4 weeks, 3 mths, 6 mths, 9 mths and one year
  Not Working, Part Time, Full Time, Retired
Visual Analog Scale (VAS) | Baseline and then Assess Changes Post Intervention at 4 weeks, 3 mths, 6 mths, 9 mths and one year
  Assesses pain based on a scale from 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Stem Cell Institute, Encino, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within six months of study completion.
Access Criteria: Solutions IRB is overseeing the study and will review data access requests.

REFERENCES:
- [Result] Aagaard-Tillery KM, Silver R, Dalton J. Immunology of normal pregnancy. Semin Fetal Neonatal Med. 2006 Oct;11(5):279-95. doi: 10.1016/j.siny.2006.04.003. Epub 2006 Jun 19. PMID 16784908
- [Result] Shay E, Kheirkhah A, Liang L, Sheha H, Gregory DG, Tseng SC. Amniotic membrane transplantation as a new therapy for the acute ocular manifestations of Stevens-Johnson syndrome and toxic epidermal necrolysis. Surv Ophthalmol. 2009 Nov-Dec;54(6):686-96. doi: 10.1016/j.survophthal.2009.03.004. Epub 2009 Aug 21. PMID 19699503
- [Result] Delo DM, De Coppi P, Bartsch G Jr, Atala A. Amniotic fluid and placental stem cells. Methods Enzymol. 2006;419:426-38. doi: 10.1016/S0076-6879(06)19017-5. PMID 17141065
- [Result] Soncini M, Vertua E, Gibelli L, Zorzi F, Denegri M, Albertini A, Wengler GS, Parolini O. Isolation and characterization of mesenchymal cells from human fetal membranes. J Tissue Eng Regen Med. 2007 Jul-Aug;1(4):296-305. doi: 10.1002/term.40. PMID 18038420
- [Result] De Coppi P, Bartsch G Jr, Siddiqui MM, Xu T, Santos CC, Perin L, Mostoslavsky G, Serre AC, Snyder EY, Yoo JJ, Furth ME, Soker S, Atala A. Isolation of amniotic stem cell lines with potential for therapy. Nat Biotechnol. 2007 Jan;25(1):100-6. doi: 10.1038/nbt1274. Epub 2007 Jan 7. PMID 17206138

DOCUMENTS (1):
  • Informed Consent Form (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03390920/ICF_000.pdf